CLINICAL TRIAL: NCT03759067
Title: Prospective Partially Randomized Comparison of Clopidogrel Loading Versus Maintenance Dosing to Prevent Periprocedural Myocardial Infarction After Stenting for a Stable Angina Pectoris
Brief Title: Method of Clopidogrel Pre-treatment Undergoing Conventional Coronary Angiogram in Angina Patients
Acronym: MECCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Do-sun Lim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUMC_MECCA
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Angina, Stable
Keywords: clopidogrel loading; maintenance dose; periprocedural MI
MeSH Terms: conditions — Angina, Stable | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LD group (Active Comparator): clopidogrel 600 mg once loading, usually 2-24 h before the procedure
  Interventions: Drug: clopidogrel 600mg
- MD group (Experimental): After randomization, the routine therapy using daily clopidogrel 75mg
  Interventions: Drug: clopidogrel 75mg
- RL group (Active Comparator): After randomization, additional clopidogrel 300 mg reloading for patients who were taking a maintenance dose.
  Interventions: Drug: clopidogrel 75mg; Drug: Clopidogrel 300 mg

INTERVENTIONS:
Drug: clopidogrel 75mg — clopidogrel once daily 75mg
  Other Names: MD
  Arms: MD group; RL group
Drug: Clopidogrel 300 mg — clopidogrel 300mg reloading
  Other Names: RL
  Arms: RL group
Drug: clopidogrel 600mg — clopidogrel 600mg loading
  Other Names: LD
  Arms: LD group

SUMMARY:
The study included 511 patients who underwent PCI because of angina during 2010-2011 at three Korean hospitals. Clopidogrel-naïve patients received either a loading dose (LD; 600 mg at 2-24 h before the procedure) or routine maintenance therapy (75 mg/day for ≥5 days) plus either a 300-mg reload (RL) or only the maintenance dose (MD).

DETAILED DESCRIPTION:
Elevation of myocardial infarction markers after coronary stenting reflects periprocedural myonecrosis or periprocedural myocardial infarction (PMI), which is associated with an increase in cardiac events and mortality. Thus, we aimed to evaluate various clopidogrel pre-treatment methods for preventing PMI among patients undergoing conventional CAG for stable angina pectoris. The Method of Clopidogrel Pre-treatment Undergoing Conventional Coronary Angiogram in Angina patients (MECCA) study was a prospective, partially randomized, multi-center clinical trial. Between October 2010 and July 2011, 511 patients underwent PCI for angina pectoris at the Korean University Anam Hospital, the Eulji Hospital, and the Hanil General Hospital. Clopidogrel-naïve patients were enrolled to receive a loading dose (the LD group; clopidogrel at 600 mg, usually 2-24 h before the procedure) or routine therapy using daily clopidogrel doses (75 mg/day for ≥5 days). Patients receiving daily doses were randomized to receive either an additional 300-mg reload (the RL group) or no additional loading (the maintenance dose [MD] group). The 600-mg or 75-mg treatment regimens were selected at the physician's discretion. The primary outcome was creatinine kinase myocardial band (CK-MB) levels at several time points. The CK-MB levels were measured at baseline, 8 h, and 24 h, while troponin-I levels were measured at 8 h after the PCI.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and, stable angina pectoris and, at least 1 ischemic evidence below

  1. Treadmil test positive
  2. ST-T change in resting ECG or 24-hour ECG
  3. Regional wall motion abnormality in Echocardiography or cardiac MRI
  4. Myocardial ischemia at MIBI scan
  5. moderate to severe stenosis at coronary CT angiography
  6. chest pain or dyspnea

Exclusion Criteria:

* AST or ALT > 3 times upper normal limits
* Serum creatinine > 2.0 mg/dL
* chronic malaborption status (disorder or operation)
* planned surgery within 1 year
* pregnancy or breast-feeding patients
* life expectancy < 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2010-10-18 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
8hour mean CK-MB | 8hour after PCI
  mean CK-MB(creatinine kinase myocardial band) is checked 8hour after PCI
24hour mean CK-MB | 24hour after PCI
  mean CK-MB(creatinine kinase myocardial band) is checked 8hour after PCI

SECONDARY OUTCOMES:
8hour mean troponin-I | 8hour after PCI
  mean troponin-I is checked 8hour after PCI
Prevalence of periprocedural myocardial infarction (PMI) | 8hour or 24hour after PCI
  Patients were considered to have PMI when their CK-MB level was elevated to >3 times the upper limit of normal, which was defined as 4.94 ng/mL.
All cause death | 9 months after PCI
  All death is evaluated using chart reviews and telephone calls.
Coronary revascularization | 9 months after PCI
  Coronary revascularization is evaluated using chart reviews and telephone. calls.

OTHER OUTCOMES:
Moderate to severe GUSTO bleeding | within 1week after PCI
  Moderate GUSTO bleeding is defined as bleeding that requires blood transfusion but does not result in hemodynamic compromise. severe GUSTO bleeding is defined as a intracranial hemorrhage or hemodynamic compromise requiring treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242